CLINICAL TRIAL: NCT01051726
Title: Effects of Aromatherapy on Childbirth
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 10018
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Parturition; Natural Childbirth; Labor Pain
Keywords: aromatherapy; childbirth; Obstetrics; Labour; Complementary Medicine; delivery, obstetric
MeSH Terms: conditions — Labor Pain | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aromatherapy group 1 (Experimental): Participants will be given essential oil consisting of (Peppermint, Lavender, Clary Sage and Frankincense) together with a swab to put the oil on.
  Interventions: Other: Aromatherapy oil
- Control group 2 (Placebo Comparator): Participants receive a bottle of non essential oil and a swab.
  Interventions: Other: None essential oil
- Control group 3 (No Intervention): Standard maternity care to measure baseline.

INTERVENTIONS:
Other: Aromatherapy oil — Oil consists of Clary Sage, Peppermint, Lavender and Frankincense with drops of each mixed into a carrier oil.
  Arms: Aromatherapy group 1
Other: None essential oil — Baby oil
  Arms: Control group 2

SUMMARY:
Aromatherapy is a form of complementary medicine that uses scented materials known as essential oils for the purpose of affecting a person's health or mood. Although aromatherapy has been used in childbirth for centuries, there are no high-quality studies examining whether the treatment works.

Methodology

We would like to see if aromatherapy affects a woman's experience of childbirth by lowering associated anxiety and pain. Consenting participants will be randomly allocated to one of these groups:

1. Aromatherapy oils (e.g. clary sage, peppermint, lavender, frankincense)
2. Non-essential oil (baby oil)
3. Standard maternity care

We will gather primary data, e.g. if she's been in labour before and her awareness of complementary medicine. We will also conduct the Spielberger State-Trait Anxiety Inventory with her, and provide her with the oil and swab if she is in groups 1 or 2 with instructions to keep the swab with the oil on it near to her. She can also put more oil on the swab as she requires.

Postnatally, data will be collected from her notes regarding pain relief used, duration of labour, augmentation of labour, and any other medical interventions of note. We will also complete the anxiety scale with her once more. Before her discharge we ask the mother for any comments regarding her experience of the labour. The results from all three cohorts will then be compared. There will also be opportunity for the midwife to make any comments regarding his/her perception of the participant's labour. Finally we will hold a focus group with midwives regarding the practicalities for implementation of aromatherapy in maternity care

ELIGIBILITY:
Inclusion Criteria:

* women in labour and expecting a normal delivery,
* aged > 16 who are able to make informed consent;
* singleton pregnancy;
* spontaneous or induced labour onset;
* prior to elective or emergency caesarean section.

Exclusion Criteria:

* preterm labour;
* pool births;
* scheduled caesarean section.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Whether aromatherapy can lower levels of anxiety in women in labour | 1 year

SECONDARY OUTCOMES:
Whether aromatherapy decreases analgesia use in women in labour | 1 year
Whether aromatherapy increases her perceived quality and satisfaction of women in labour | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dawn-Marie Walker, BSc MSc PhD, Principal Investigator — University of Nottingham
Locations (1):
- Kings Mill Hospital, Nottingham, United Kingdom